CLINICAL TRIAL: NCT01547000
Title: Guanfacine in Children With Tic Disorders: A Multi-site Study
Brief Title: Guanfacine in Children With Tic Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); University of South Florida (Other); Shire (Industry); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1004006635
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Tourette Disorder; Tourette Syndrome
Keywords: Tourette Syndrome; Tourette Disorder; Tics; Motor tics; Vocal tics; Intuniv; Guanfacine; Medication; Drug; Placebo; Child; Children; Adolescent
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inactive placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Extended-release Guanfacine (Experimental)
  Interventions: Drug: extended-release guanfacine (Intuniv)

INTERVENTIONS:
Drug: placebo — Administered up to 8 weeks.
  Arms: Inactive placebo
Drug: extended-release guanfacine (Intuniv) — 1 mg tablets; flexible dosing up to 4 mg/day for up to 16 weeks.
  Other Names: Intuniv
  Arms: Extended-release Guanfacine

SUMMARY:
The goal of this pilot study is to obtain preliminary information on the tolerability and efficacy of extended release guanfacine (trade name Intuniv) in children with Tourette Disorder (TD, also called Tourette syndrome).

DETAILED DESCRIPTION:
Guanfacine is commonly used for the treatment of tics in children with Tourette Disorder, but neither the immediate release compound nor the new extended release formulation have been evaluated for tics as a primary outcome. This pilot study is not designed to demonstrate efficacy of extended release guanfacine in the treatment of tics in children with TD. Rather, the goal of this trial is to determine whether extended release guanfacine warrants further study in a large scale trial. Immediate-release guanfacine is frequently used in children with TD, but dosing, time to effect and adverse effects with the new extended release guanfacine are unknown. The use of placebo in this trial reduces bias in the measurement of outcomes because it ensures blindness in the parent and clinician ratings.

This is a three-site, investigator-initiated, randomized, double-blind, placebo-controlled, parallel-group study. Subjects who show a positive response to extended release guanfacine in the 8-week double-blind phase will continue on the the drug in an 8-week extension phase. Subjects who are randomly assigned to placebo and do not show improvement will be offered 8-weeks of open-label treatment with Intuniv.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tourette Disorder or chronic motor or vocal tic disorder.
* Between ages 6 yrs 0 mos and 17 years 0 months.
* Weight >/= 15 kg (33 lbs).
* Ability to swallow pills whole.

Exclusion Criteria:

* IQ < 80.
* Positive pregnancy test.
* Positive drug test.
* Low blood pressure.
* Prior history of hypersensitivity to guanfacine.
* Prior failed treatment with an adequate trial of guanfacine in last 2 years.
* Concurrent treatment with another psychoactive medication for tics, stimulant medication, or Habit Reversal therapy.
* Medication for OCD, anxiety or depression will be allowed if dose is stable for 8 wks with no planned changes; SSRIs are allowed.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D Scahill, MSN, PhD, Study Director — Emory University; Barbara J Coffey, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai; Tanya Murphy, MD, MS, Principal Investigator — University of South Florida; Thomas Fernandez, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale Child Study Center, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Mount Sinai School of Medicine, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inactive Placebo | Extended-release Guanfacine
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactive Placebo | Extended-release Guanfacine | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 16 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.2) | 11.5 (11) | 11.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Tanner stage [Count of Participants; unit: Participants] — The Tanner scale categorizes physical measurements of development based on external primary and secondary sex characteristics, such as the size of the breasts, genitals, testicular volume and development of pubic hair in children, adolescents, and adults. There is insufficient space given in this form to list all of the measurements here. In brief, Stage 1: no pubic hair; Stage 2: initial growth of pubic hair, breasts, nipples, scrotum, testes; Stage 3: additional growth of all mentioned in Stage 2.
  Participants
    Stage 1 or 2 | 11 | 10 | 21
    Stage 3+ | 7 | 6 | 13
Yale Global Tic Severity Scale (YGTSS) [Mean (Standard Deviation); unit: units on a scale] — The YGTSS is a clinician-rated scale that begins with a systematic inquiry of tic symptoms in the preceding week. Current motor and phonic tics are rated separately according to number, frequency, intensity, complexity, and interference, each rated on 0 to 5 scale with higher scores indicating greater severity/worse outcome (Leckman et al. 1989). The YGTSS yields a total motor score (0-25), a total phonic score (0-25), a total tic score (sum of total motor and total phonic scores; 0-50), and an impairment score (0-50). Higher scores indicate greater severity/worse outcome.
  units on a scale
    Total Tic Score | 27.7 (8.7) | 26.3 (6.61) | 27.0 (10.9)
    Total Motor score | 17.2 (3.44) | 15.2 (2.61) | 16.3 (4.3)
    Total Phonic score | 10.4 (6.73) | 11.1 (6.13) | 10.7 (9.1)
    Impairment | 28.6 (8.01) | 29.8 (8.18) | 29.2 (11.4)
Clinical Global Impressions (CGI) [Count of Participants; unit: Participants]
  Moderately ill | 9 | 12 | 21
  Markedly ill | 6 | 4 | 10
  Severely ill | 3 | 0 | 3
Tic Symptom Self-Report (TSSR) [Mean (Standard Deviation); unit: units on a scale] — The TSSR (Cohen and Leckman 1984) was completed by a parent or caretaker. It includes 20 motor and 20 phonic tics, each rated 0 to 3. The motor and phonic scores are summed to create a total score. The total score for Tic Symptom Self-Report ranged from 0-120. Higher scores means greater severity/worse outcome. It has been shown to be sensitive to treatment effects (Scahill et al. 2003).
  units on a scale | 24.6 (16.94) | 26.9 (22.83) | 25.7 (28.5)
Premonitory Urge for Tics Scale (PUTS) [Mean (Standard Deviation); unit: units on a scale] — The PUTS (Woods et al. 2005) is a 10-item self-report measure of premonitory urges in individuals with tics. Individual item scores (1-4) are summed, yielding a total score (10-40) reflecting the presence and frequency of pre-tic (i.e., premonitory) urges along with relief that may be experienced after tics have been completed. Higher scores means higher frequency of premonitory urges.
  units on a scale | 20.9 (8.18) | 19.8 (5.39) | 20.4 (9.8)
Attention-Deficit/Hyperactivity Disorder Rating Scale (parent) [Mean (Standard Deviation); unit: units on a scale] — The ADHD Rating Scale (Reid et al. 1998) is an 18-item, DSM-IV referenced measure rated by a parent or caretaker in this study. The sum of nine inattention items and nine hyperactivity/impulsiveness items (each rated on a 0-3 scale) are included in the total score. The total score for the Attention-Deficit/Hyperactivity Disorder Rating Scale (parent) ranged from 0 to 54. A higher score means greater severity of ADHD symptoms.
  units on a scale | 17.5 (13.65) | 19.7 (12.29) | 18.5 (18.4)
Disruptive Behavior Rating Scale (DBRS) [Mean (Standard Deviation); unit: units on a scale] — The DBRS (Barkley and Murphy 2006) is an 8-item measure of oppositional defiant disorder rated by the parent or caretaker, with each item rated on a 0 to 3 scale. The total score is the sum of all 8 item scores. The total score for the Disruptive Behavior Rating Scale (DBRS) ranged from 0 to 24. Higher scores means greater severity of disruptive behaviors. Scores of 12 and higher are considered clinically significant.
  units on a scale | 5.6 (7.37) | 8.8 (6.59) | 7.1 (9.9)
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) [Mean (Standard Deviation); unit: units on a scale] — The CY-BOCS (Scahill et al. 1997) is a 10-item, semistructured interview administered by the independent evaluator and is designed to rate the severity of obsessive-compulsive disorder. Scores range from 0 to 40 with higher scores indicating greater severity.
  units on a scale | 10.5 (11.43) | 9.6 (10.41) | 10.1 (15.5)
Rage Outbursts and Anger Rating Scale (ROARS) [Mean (Standard Deviation); unit: units on a scale] — The ROARS (Budman et al. 2008) is a 3-item, clinician-rated scale designed to quantify the severity of explosive outbursts in the past week, administered by an independent evaluator. The items are rated from 0 to 3 on frequency, intensity, and duration and then added together for a total score. The total score for the Rage Outbursts and Anger Rating Scale (ROARS) ranged from 0 to 9. Higher scores indicates greater severity.
  units on a scale | 2.2 (2.87) | 3.1 (2.87) | 2.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Yale Global Tic Severity Scale (YGTSS)
Description: The YGTSS is a clinician-rated scale that begins with a systematic inquiry of tic symptoms in the preceding week. Current motor and phonic tics are rated separately according to number, frequency, intensity, complexity, and interference, each rated on 0 to 5 scale with higher scores indicating greater severity/worse outcome (Leckman et al. 1989). The YGTSS yields a total motor score (0-25), a total phonic score (0-25), a total tic score (sum of total motor and total phonic scores; 0-50), and an impairment score (0-50). Higher scores indicate greater severity/worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactive Placebo | Extended-release Guanfacine
Number analyzed (Participants) | 18 | 16
units on a scale
  Total tic score | 24.72 (10.54) | 23.56 (6.42)
  Total Motor score | 15.00 (5.87) | 12.94 (3.43)
  Total Phonic Score | 9.72 (6.43) | 10.63 (5.49)
  Impairment | 23.44 (11.51) | 26.44 (9.61)

ADVERSE EVENTS:
Arm/Group | Inactive Placebo | Extended-release Guanfacine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/16
Other Adverse Events (participants affected / at risk) | 4/18 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inactive Placebo (N=18) | Extended-release Guanfacine (N=16)
depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inactive Placebo (N=18) | Extended-release Guanfacine (N=16)
Fatigue/tiredness (General disorders) | 3 | 14
Drowsiness (General disorders) | 3 | 12
Dry mouth (General disorders) | 4 | 10
Headache (General disorders) | 2 | 10
Irritability (Social circumstances) | 1 | 9
Stomach ache (Gastrointestinal disorders) | 2 | 8
Decreased appetite (General disorders) | 3 | 8
Depressed mood (Psychiatric disorders) | 1 | 7
Dizziness (General disorders) | 1 | 7
Emotional/tearful (General disorders) | 4 | 6
Daydreaming (General disorders) | 2 | 6
Trouble falling asleep (General disorders) | 4 | 5
Hypotension (Cardiac disorders) | 1 | 3
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 3
Other vision problems (Eye disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 4 | 2
Mid-sleep awakening (General disorders) | 3 | 2
Increased energy (General disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Increased appetite (General disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
We are limited by the small size of this subgroup to determine whether children with comorbid CTD and ADHD might have a significant response to extended-release guanfacine, both with regard to tics and ADHD symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No